CLINICAL TRIAL: NCT04346797
Title: CORIMUNO19-ECU: Trial Evaluating Efficacy and Safety of Eculizumab (Soliris) in Patients With COVID-19 Infection, Nested in the CORIMUNO-19 Cohort
Acronym: CORIMUNO19-ECU
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200375-4
Record Dates: First submitted 2020-04-06; First posted 2020-04-15 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: SARS-CoV-2; COVID19
MeSH Terms: conditions — COVID-19 | interventions — eculizumab

STUDY DESIGN:
Intervention Model Description: Bayesian open labelled randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eculizumab (Experimental): Eculizumab
  Interventions: Drug: Eculizumab
- Standard of Care (No Intervention): Best standard of care

INTERVENTIONS:
Drug: Eculizumab — Intravenous administration as follows:
  Induction dosage regimen at 1200 mg on Days 1, 4, 8 then 1200 mg or 900 mg on Day 12 depending on the monitoring of Eculizumab Plasma Level and CH5O and sC5B9 and maintenance doses of 900 mg on Days 15, 18 and 22
  Arms: Eculizumab

SUMMARY:
The overall objective of the study is to determine the therapeutic effect and tolerance of Eculizumab in patients with moderate, severe pneumonia or critical pneumonia associated with Coronavirus disease 2019 (COVID-19). Eculizumab is a terminal complement inhibitor that has been investigated for more than 10 years in numerous complement-mediated diseases. The study has a cohort multiple Randomized Controlled Trials (cmRCT) design. Randomization will occur prior to offering Eculizumab administration to patients enrolled in the CORIMUNO-19 cohort. Eculizumab will be administered to consenting adult patients hospitalized with COVID-19 either diagnosed with moderate or severe pneumonia requiring no mechanical ventilation or critical pneumonia requiring mechanical ventilation. Patients who will chose not to receive Eculizumab will receive standard of care. Outcomes of Eculizumab-treated patients will be compared with outcomes of standard of care-treated patients as well as with outcomes of patients treated with other immune modulators.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 675 years old included in the CORIMUNO-19 cohort
2. Patients belonging to one of the 2 following groups

   * Group 1: 60 patients not requiring ICU at admission with moderate and severe pneumopathy according to the WHO Criteria of severity of COVID pneumopathy, meeting all of the 2 following criteria:

     * Respiratory symptoms with radiological findings of pneumonia
     * Severe pneumonia requiring ≥ 5L/min of oxygen to maintain SpO2 >97%
   * Group 2: 60 patients requiring ICU based on Criteria of severity of COVID pneumopathy.

     * Respiratory failure and requiring mechanical ventilation
     * Vasopressive support
3. Vaccinated against meningococcal infections within 3 years prior to, or at the time of, initiating Eculizumab to reduce the risk of meningococcal infection (N meningitidis) [(Bexsero® (2 injections with a minimum of 1 month interval) + Menveo@ or Niminrex® ) and daily antibiotics (Oracilline®)]. If vaccination cannot be confirmed or if the patient cannot receive it, the participant should receive prophylactic antibiotics against meningococcal infection prior to initiating Eculizumab treatment and for at least 3 months from the last infusion of Eculizumab.
4. Female patients of childbearing potential and male patients with female partners of childbearing potential must follow protocol-specified guidance for avoiding pregnancy while on treatment and for 8 months after last dose of Eculizumab.

5- Body weight ≥40 kg

6-Patient and/or alternatively by next-of-kin must be willing and able to give written informed consent according to the applicable regulations including emergency and intensive care contexts

Exclusion Criteria:

* Patients with exclusion criteria to the CORIMUNO-19 cohort.
* Age ≥ 70 years
* Pregnancy or lactation
* History or unresolved Neisseria meningiditis infection
* Ongoing sepsis, presence or suspicion of active and untreated systemic bacterial infection prior study screening and untreated with antibiotics,
* Hypersensitivity to any ingredient contained in Eculizumab, including hypersensitivity to murine proteins.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival without needs of intubation at day 14 | 14 days
  Survival without needs of intubation, events considered are intubation or death
Change in organ failure at day 3 | 3 days
  Change in organ failure at day 3, defined by the relative variation in Sequential Organ Failure Assessment score

SECONDARY OUTCOMES:
Intubation free survival at day 14 | Day 14
  Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by NIV or High flow: 6 Intubation and Mechanical ventilation, pO2/FIO2>=150 OR SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO: 9 Dead: 10
WHO progression scale at days 4, 7 and 14 | 4, 7 and 14 days
  WHO progression scale:
  Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by NIV or High flow: 6 Intubation and Mechanical ventilation, pO2/FIO2>=150 OR SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO: 9 Dead: 10
Survival at 14, 28 and 90 days | 14, 28 and 90 days
  Overall survival
Time to discharge | 90 days
  Time between inclusion and hospital discharge
Time to oxygen supply independency | 90 days
  Time between inclusion and oxygen supply independency
Time to negative viral excretion | 90 days
  Time between inclusion and negative viral excretion
Incidence of secondary infections | 90 days
  Incidence of secondary infections (acquired pneumonia)
Vasopressor-free survival | 90 days
  Vasopressor-free survival
Ventilator-free survival | 90 days
  Ventilator-free survival
28-day ventilator-free days | 28 days
  Number of ventilator-free days alive up to day 28
Incidence of dialysis | 90 days
  Incidence of dialysis (renal replacement therapy)
PaO2/FiO2 ratio | days 4, 7, 14
  PaO2/FiO2 ratio
Rate of respiratory acidosis at day 4 | 4 days
  Number of patients with arterial blood pH of <7.25, with a partial pressure of arterial carbon dioxide [Paco2] of ≥60 mm Hg for >6 hours
Time to ICU discharge | 90 days
  Time to ICU discharge

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Réanimation médicale, Paris
  - saint Louis, Paris
  - Saint Louis, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided